CLINICAL TRIAL: NCT00000231
Title: Buprenorphine Detoxification With Two Types of Treatment. BBD IV
Brief Title: Buprenorphine Detoxification With Two Types of Treatment. BBD IV - 13
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-13; R01-06969-13
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1994-03

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate buprenorphine and behavioral treatment with and without contingent payment on compliance with pro-social activities. In addition, we will examine whether blind naltrexone dosing is effective in indicating naltrexone consumption.

ELIGIBILITY:
Please contact site for information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1992-02

PRIMARY OUTCOMES:
Drug use
Retention
Weeks abstinent
Weeks continuous abstinence
Overall treatment outcome
Naltrexone consumption

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Derived] Bunyoz KI, Tsikandylakis G, Mortensen K, Gromov K, Mohaddes M, Malchau H, Troelsen A. No difference in whole-blood metal ions between 32-mm and 36- to 44-mm femoral heads in metal-on-polyethylene total hip arthroplasty: a 2-year report from a randomised control trial. Hip Int. 2023 Mar;33(2):184-192. doi: 10.1177/11207000211022623. Epub 2021 Jun 8. PMID 34102902